CLINICAL TRIAL: NCT00583349
Title: A Combined Phase I and Phase II Trial of Intravesical Abraxane, a Biologically Interactive Albumin-bound Paclitaxel, in the Treatment of Refractory Non-muscle Invasive and in T2 Transitional Cell Bladder Cancer
Brief Title: Intravesicular Abraxane for Treatment-Refractory Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAC1114
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Chemotherapy; Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abraxane administration (Experimental): Phase I and Phase II: Patients will receive intravesical Abraxane by sterile urethral catheterization once weekly for six weeks.
  Phase II: If a complete response after six weekly installations is achieved, patients will receive additional monthly maintenance instillations until there is a positive cystoscopic biopsy or until a maximum of six additional instillations have been administered.
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — Abraxane is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug.
  Intravesically administered, dose escalation, 6 weekly instillations
  Other Names: Paclitaxel protein-bound

SUMMARY:
Phase I:

To determine the safety, toxicity and efficacy profiles of intravesically administered Abraxane at the Maximum Tolerated Dose.

To assemble tissue bank to assess molecular correlates for response to intravesical Abraxane therapy. The antibodies analyzed will include p53, p63, Stathmin, Tau and Ki67.

Phase II:

To evaluate the utility (potential for clinical efficacy) of Abraxane in the treatment of refractory non-muscle invasive and a subset of T2 TCC of the bladder as measured by response rate (defined as negative cytology and bladder biopsy).

To further evaluate the safety and toxicity profile of intravesically administered Abraxane therapy.

DETAILED DESCRIPTION:
In 2006, it is estimated that 61,420 cases of bladder cancer will be diagnosed in the United States and 13,060 people will die from the disease. This makes bladder cancer the fourth leading cause of cancer in men and the ninth leading cause of cancer in women in the United States. Non-muscle invasive bladder cancer accounts for 70 to 80 percent of these cases and the natural history can vary widely with recurrence being common. In individual cases with high-risk clinical and pathological features (Ta, Tis, and T1) the use of intravesical therapy following complete transurethral resection of the tumor has become the standard of care. However up to 50 percent of patients treated with intravesical therapy for high-risk non-muscle invasive bladder cancer will recur. Response rates to second-line intravesical therapy are 20 percent or less in this population. Innovations in the efficacy of intravesical agents also have applications within a subset of patients with muscle-invasive disease who are undergoing complete transurethral resection in conjunction with local chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of transitional cell carcinoma (TCC) of the urinary bladder confirmed at the study institution. The patient must have demonstrated superficial recurrent bladder cancer refractory to standard intravesical therapy. This will include stage Ta, T1, Tis and exclude all patients with muscle invasion (T2). All patients with stage Ta will require documentation of high-grade histology. All grossly visible disease must be fully resected and pathologic stage will be confirmed at the institution where the patient is enrolled. Patients must exhibit disease recurrence after receiving some form of standard intravesical therapy, including Bacillus Calmette-Guerin (BCG), mitomycin, interferon or any combination thereof.
* Age > 18 and must be able to read, understand and sign informed consent
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0,1 (See Appendix II )
* Peripheral neuropathy: must be < grade 1
* Hematologic-Inclusion within 2 weeks of start of treatment

  * Absolute neutrophil count > 1,500/mm3
  * Hemoglobin >9.0 g/dl
  * Platelet count > 100,000/mm3
* Hepatic-Inclusion within 2 weeks of entry

  * Total Bilirubin must be within normal limits.
  * Adequate renal function with serum creatinine ≤ 2.0 mg/dL
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) for the institution, Alkaline phosphatase ≤ 2.5 x ULN for the institution, unless bone metastasis is present in the absence of liver metastasis
* Women of childbearing potential must have a negative pregnancy test.
* All patients of childbearing potential must be willing to consent to using effective contraception, i.e., intrauterine device (IUD), Birth control pills, Depo-Provera, and condoms while on treatment and for 3 months after their participation in the study ends.
* No intravesical therapy within 6 weeks of study entry
* No prior radiation to the pelvis

Exclusion Criteria:

* Prior systemic docetaxel or paclitaxel therapy.
* Any other malignancy diagnosed within 2 years of study entry (except basal or squamous cell skin cancers or non-invasive cancer of the cervix) is excluded.
* Concurrent treatment with any chemotherapeutic agent.
* Women who are pregnant or lactating.
* History of vesicoureteral reflux or an indwelling urinary stent.
* Participation in any other research protocol involving administration of an investigational agent within 3 months prior to study entry aside from the phase I segment of this study.
* History of neuropathy of any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M McKiernan, MD, Principal Investigator — Columbia University Irving Medical Center, Urology
Locations (1):
- Herbert Irving Pavillion 11th Floor, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Abraxane 150 mg: Phase 1, dose level 1: Patients will receive intravesical 150 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 225 mg: Phase 1, dose level 2: Patients will receive intravesical 225 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 300 mg: Phase 1, dose level 3: Patients will receive intravesical 300 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 375 mg: Phase 1, dose level 4: Patients will receive intravesical 375 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 450 mg: Phase 1, dose level 5: Patients will receive intravesical 450 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 500 mg: Phase 1, dose level 6: Patients will receive intravesical 500 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- MTD: Abraxane 500 mg: Phase 2: Patients will receive the maximum tolerated dose (MTD) intravesical 500 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
Period: Phase 1: Dose Level 1
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 2
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 0 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 3
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 4
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 0 | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 5
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 0 | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 0 | 0
Period: Phase 1: Dose Level 6
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 0 | 0 | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: Maximum Tolerated Dose
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 28 | 46
Age, Customized [Count of Participants; unit: Participants]
  ≥ 18 years | 3 | 3 | 3 | 3 | 3 | 3 | 28 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 1 | 1 | 6 | 11
  Male | 3 | 2 | 2 | 2 | 2 | 2 | 22 | 35
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 28 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: To determine the safety, toxicity and efficacy profiles of intravesically administered Abraxane at the Maximum Tolerated Dose (MTD). A DLT is defined by the National Cancer Institute Common Toxicity Criteria version 3.0
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Abraxane 150 mg: Phase 1, dose 1: Patients will receive intravesical 150 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 225 mg: Phase 1, dose 2: Patients will receive intravesical 225 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 300 mg: Phase 1, dose 3: Patients will receive intravesical 300 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 375 mg: Phase 1, dose 4: Patients will receive intravesical 375 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 450 mg: Phase 1, dose 5: Patients will receive intravesical 450 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 500 mg: Phase 1, dose 6: Patients will receive intravesical 500 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 28
Participants
  Grade 1 local toxicity | 2 | 2 | 1 | 3 | 0 | 3 | 4
  Grade 2 local toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Grade 3 or higher local toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Complete Response (CR) or No Response (NR) After Treatment
Description: To evaluate the utility (potential for clinical efficacy) of Abraxane in the treatment of refractory superficial transitional cell carcinomas (TCC) as measured by response rate (defined as negative cytology and bladder biopsy). Patients were considered to have a complete response if they had a negative biopsy and negative cytology. All patients with positive biopsies or cytology were classified as having no response.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 28
participants
  CR | 1 | 3 | 0 | 1 | 0 | 0 | 10
  NR | 2 | 0 | 3 | 2 | 3 | 3 | 18

3. Secondary Outcome: To Further Evaluate the Safety and Toxicity Profile of Intravesically Administered Abraxane Therapy.
Time Frame: 6 months
Population: Data were not collected.
Groups:
- Abraxane Administration: Patients will restrict their fluid intakes the morning of treatments and will have emptied their bladders at each of their visits and have up to 100ml of Abraxane solution administered to their bladder via urinary catheter once weekly for six weeks.
  Paclitaxel, nanoparticle albumin-bound: Intravesically administered, dose escalation, 6 weekly instillations
Arm/Group | Abraxane Administration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Abraxane 150 mg; Abraxane 225 mg: Patients will receive intravesical 150 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 300 mg: Patients will receive intravesical 300 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 375 mg: Patients will receive intravesical 375 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 450 mg: Patients will receive intravesical 450 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
- Abraxane 500 mg: Patients will receive intravesical 500 mg Abraxane by sterile urethral catheterization once weekly for six weeks.
Arm/Group | Abraxane 150 mg | Abraxane 225 mg | Abraxane 300 mg | Abraxane 375 mg | Abraxane 450 mg | Abraxane 500 mg | MTD: Abraxane 500 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 2/28
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/28
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 2/3 | 1/3 | 2/3 | 1/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane 150 mg (N=3) | Abraxane 225 mg (N=3) | Abraxane 300 mg (N=3) | Abraxane 375 mg (N=3) | Abraxane 450 mg (N=3) | Abraxane 500 mg (N=3) | MTD: Abraxane 500 mg (N=28)
Systemic Absorption of Drug (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 — 1 subject had detectable systemic absorption of the drug after 1 instillation of the 450 mg dose (level 16 ng/ml). Instillation was delayed by 1 week, after which serum levels returned to undetectable and remained so for the remainder of treatment.
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No